CLINICAL TRIAL: NCT06413628
Title: Efficiency of Different Treatment Modalities on Radiation Induced Trismus for Maxillofacial Cases
Brief Title: Efficiency of Different Treatment Modalities on Radiation Induced Trismus for Maxillofacial Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: A02011023RP
Record Dates: First submitted 2024-03-19; First posted 2024-05-14 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-03

CONDITIONS: Trismus; Cancer
MeSH Terms: conditions — Trismus; Neoplasms | interventions — Low-Level Light Therapy

STUDY DESIGN:
Intervention Model Description: group I received threaded tapered screw appliance therapy , patients in group II received low-level laser therapy, and patients in group III received low-level laser therapy in addition to threaded tapered screw appliance therapy.
Who Masked: Investigator
Masking Description: The randomization and assignment of patients to treatment groups was carried out by dental experts who were not informed about the treatment groups.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- threaded tapered screw appliance therapy (Active Comparator): The appliance was digitally designed by solid works programs for 3rd CAD design software to obtain the STL file format. The virtual design of was approved. The printer was loaded with material of 3D-printed denture base. The appliance was printed.
  Interventions: Other: screw tapered appliance
- low-level laser therapy (Active Comparator): The laser apparatus consisted of a handpiece with two attachments: either a plastic tip was attached to the same handpiece to transfer laser energy intra-orally when it was used to irradiate the lateral pterygoid muscle, or a specially designed optic prism was attached to the tip of the prism for extraoral application on extraoral muscles.
  Interventions: Other: screw tapered appliance
- low level laser therapy combined with appliance (Active Comparator): low-level laser therapy in addition to threaded tapered screw appliance therapy as mentioned previously in group I and group II
  Interventions: Other: screw tapered appliance

INTERVENTIONS:
Other: screw tapered appliance — The appliance was digitally designed by solid works programs for 3rd CAD design software to obtain the STL file format. The virtual design of was approved. The printerwas loaded with material of 3D-printed denture base. The appliance was printed.
  Other Names: low level laser therapy

SUMMARY:
Aim: to compare different treatment modalities for radiation induced trismus for maxillofacial patients methods:45 participants (20 females and 25 males) with trismus and pain following head and neck cancer and underwent radiation therapy were enrolled in this study . patients were divided into three groups : group1 received threaded tapered screw appliance therapy, patients in group II received low-level laser therapy and patients in group III received low-level laser therapy in addition to threaded tapered screw appliance therapy.

DETAILED DESCRIPTION:
All patients received treatment according to their group: For group I, received threaded tapered screw appliance therapy . The appliance was digitally designed by solid works programs for 3rd CAD design software to obtain the STL file format. The virtual design of was approved. The printer was loaded with material of 3D-printed denture base. The appliance was printed.

For group II received low-level laser therapy, the laser type was of diode laser.The laser apparatus consisted of a hand piece with two attachments: either a plastic tip was attached to the same hand piece to transfer laser energy intro-orally when it was used to irradiate the lateral pterygoid muscle, or a specially designed optic prism was attached to the tip of the prism for extraoral application on extra oral muscles. All patients in this group received low level laser therapy twice times a week for 6 weeks totaling 12 sessions. In each session, the laser beam was applied in a three phases treatment protocol as follows: (a) The insertion of the lateral pterygoid muscle into the condylar neck and disc was treated in the first phase by applying a laser beam 1 cm anterior to the condyle below the zygomatic arch. (b) Tender spots in the masseter and temporalis muscles that were found during the initial assessment were exposed to radiation during the second phase. (c) The lateral pterygoid muscle origin was exposed to radiation in the third phase, which was performed with the mouth slightly open and intro-orally posterior to the final molar. During each phase, the laser was operated for two minutes per area at a wavelength of 810 nm and a peak output of 500 mW. It was applied continuously, a little distance away from the tissues. The laser probe was positioned perpendicular to the target area. Prior to usage, the laser was calibrated. Protective glasses were worn by the clinician and the patients. For group III, received low-level laser therapy in addition to threaded tapered screw appliance therapy as mentioned previously in group I and group II. Concurrent with the initial low level laser therapy session, screw tapered appliance was used for the first time.

Throughout the trial, no medication was administered to any of the groups. The patients were not allowed to use any painkillers or analgesics.

ELIGIBILITY:
Inclusion Criteria:

* (a) Clinical diagnosis of trismus in head and neck cancer patients who received radiation therapy
* (b) unable to chew, swallow and muscles stiffness

Exclusion Criteria:

* (a) patients with Bell's palsy
* (b) patients still receiving radiation.

Ages: 55 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2022-04-11 (Actual); Primary Completion 2022-08-13 (Actual); Study Completion 2023-12-10 (Actual)

PRIMARY OUTCOMES:
patient satisfaction(Quality of life) assessed by the Gothenburg Trismus Questionnaire (GTQ) which is a trismus-specific self-administered questionnaire | six months
  was assessed using Gothenburg trismus questionnaire witha scale ranging between 0-100, where a higher score indicates greater perceived dysfunction due to trismus. It contains three main domains 1-Jaw related problems 2- Eating limitations 3-Muscular tension
Satisfaction assessed by the (VAS)visual analogue scale of pain | six months
  the patients filled out a self-assessment 0 to 10 visual analogue scale (VAS) for Pain (where 0 equals no pain and 10 is the most severe pain)

CONTACTS AND LOCATIONS:
Overall Officials: marwa aboelez, PhD, Study Director — Mansoura University
Locations (1):
- Marwa Aboelez, Al Mansurah, Egypt

REFERENCES:
- [Result] Dijkstra PU, Huisman PM, Roodenburg JL. Criteria for trismus in head and neck oncology. Int J Oral Maxillofac Surg. 2006 Apr;35(4):337-42. doi: 10.1016/j.ijom.2005.08.001. Epub 2005 Nov 8. PMID 16280237
- [Derived] Aboelez MA, Ibrahim AM, ElSawy MA, Sayed El-Khamisy NE. Efficiency of different treatment modalities on radiation induced trismus for maxillofacial cases: a parallel randomized clinical trial. BMC Oral Health. 2025 Mar 4;25(1):332. doi: 10.1186/s12903-025-05600-7. PMID 40038715